CLINICAL TRIAL: NCT03875066
Title: Immediate Effects of Stepping Training With or Without External Feedback on Walking and Functional Ability in Ambulatory Patients With Spinal Cord Injury
Brief Title: Immediate Effects of Stepping Training Using External Feedback in Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr., Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PHD57K0194
Record Dates: First submitted 2019-03-10; First posted 2019-03-14 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-03

CONDITIONS: Spinal Cord Injuries
Keywords: Rehabilitation; Neurological condition; Walking ability; Feedback; External information
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A to B (Other): Subjects were involved in an control training program (A). After 2 weeks washout period, Subjects were trained using the other program (B).
  Interventions: Other: Stepping training without feedback; Other: Stepping training with feedback
- B to A (Other): Subjects were involved in an control training program (B). After 2 weeks washout period, Subjects were trained using the other program (A).
  Interventions: Other: Stepping training without feedback; Other: Stepping training with feedback

INTERVENTIONS:
Other: Stepping training without feedback — Subjects stand in a step standing position with placing one leg on the load cells of the device and the other leg at the posterolateral direction to the trained leg outside the load cells. Then subjects will be instructed to shift/take their body-weight onto the trained leg as most as they can. If the subjects can take a proper level of their body-weight onto the trained leg, the subjects can step the other leg forward to the marker. Then they have to do the same when steps the leg backward.
  Other Names: Control program
Other: Stepping training with feedback — Subjects stand in a step standing position with placing one leg on the load cells of the device and the other leg at the posterolateral direction to the trained leg outside the load cells, look at the displayed section which will be positioned at their eye level. Then subjects will be instructed to shift/take their body-weight onto the trained leg until the green zone of the displayed section is lightened. When the subjects can take a proper level of their body-weight onto the trained leg, the beep sound will be alarmed to trigger the subjects and therapist that the subjects can step the other leg forward to the marker. Then they have to do the same when steps the leg backward.
  Other Names: Experimental program

SUMMARY:
* Does stepping training with or without external feedback change functional ability of ambulatory patients with iSCI immediately after training?
* Are there significant differences between the immediate effects of stepping training with or without external feedback in ambulatory patients with iSCI?

DETAILED DESCRIPTION:
To compare immediate effects of stepping training with or without the utility of external feedback on functional ability relating to walking in ambulatory patients with iSCI (between-group comparison).

Secondary objective To compare immediate effects in a group of stepping training with or without the utility of external feedback on functional ability relating to walking in ambulatory patients with iSCI (within-group comparison).

ELIGIBILITY:
Inclusion Criteria:

* Independent ambulatory patients with iSCI at a chronic stage (Post-injury time > 12 months)
* Traumatic cause or non-progressive disease
* Independent walking with or without assistive devices at least 17 meters (Functional Independence Measure Locomotor (FIM-L) scores 5-7)
* Age at least 18 years
* Body mass index (BMI) between 18.5 - 29.9 kg/m2.

Exclusion Criteria:

* Any conditions or disorders that might affect ability to participate in the study and/or ambulatory ability of the subjects such as

  * Brain function disorders
  * Visual deficits that cannot be corrected using glasses or contact lens
  * Musculoskeletal pain (with an intensity of pain more than 5 out of 10 on a numerical rating pain scale)
  * Deformity of the musculoskeletal system
  * Unable to follow a command of the tests
  * Unstable medical conditions
  * Color blindness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change of walking balance using Timed up and go test [TUGT] | Baseline and immediately after complete one section training program
  The test was designed to measure mobility and dynamic balance control related to walking. Subjects will be instructed to stand up from a standard chair, walk at a fastest and safe speed for 3 meters, turn around a traffic cone, walk back and sit down on the chair with or without a walking device. Then the average time required for the 3 trials will be recorded.

SECONDARY OUTCOMES:
Change of walking speed using 10 meter walk test (10MWT) | Baseline and immediately after complete one section training program
  The test assessed the time required over the 4 m in the middle of the 10-m walkway at a comfortable and fastest speed with or without an assistive device. The time was converted to a walking speed using the formula:
  velocity (m/s) = distance (m)/ time (second).
Change of lower limb muscle strength using Five times sit-to-stand [FTSST] | Baseline and immediately after complete one section training program
  The test has used to quantify lower extremity motor strength. The time taken to complete 5 chair-rise cycles at a fastest and safe speed will be recorded for each subject. Then the average time required for the 3 trials will be used for data analysis.
Change of lower limb support ability [LLSA] on more and less affected legs | Baseline and immediately after complete one section training program
  The test was assessed to reflect a risk of musculoskeletal disorders. Participants stood upright with placing the tested leg on the digital load cell (Model L6E3-C, accuracy up to 0.1 kg, and uncertainty of the measurement ± 0.082 kg: patent application number 1701004050) and the other leg posterolaterally to the tested leg. Participants were instructed to shift their body-weight anterolaterally onto the tested leg as much as they could, and step the other leg forward, with or without using the arms according to their ability. Then the LLSA data was reported in term of percent of the participant's body-weight. These data were presented for the less and more affected limbs as identified using the sensorimotor scores. Each participant performed five trials per leg, the first two trials served as practice trials, and an other three trials were used for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, Principal Investigator — Faculty of Associated Medical Sciences, Khon Kaen University, Thailand
Locations (1):
- Faculty of Associated Medical Science, Khon Kaen, Muang, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ada L, Dean CM, Lindley R, Lloyd G. Improving community ambulation after stroke: the AMBULATE Trial. BMC Neurol. 2009 Feb 11;9:8. doi: 10.1186/1471-2377-9-8. PMID 19208261
- [Background] Amatachaya S, Amatachaya P, Keawsutthi M, Siritaratiwat W. External cues benefit walking ability of ambulatory patients with spinal cord injury. J Spinal Cord Med. 2013 Nov;36(6):638-44. doi: 10.1179/2045772312Y.0000000086. Epub 2013 Apr 12. PMID 24090447
- [Background] Amatachaya S, Keawsutthi M, Amatachaya P, Manimmanakorn N. Effects of external cues on gait performance in independent ambulatory incomplete spinal cord injury patients. Spinal Cord. 2009 Sep;47(9):668-73. doi: 10.1038/sc.2008.168. Epub 2009 Jan 13. PMID 19139759
- [Background] Amatachaya S, Naewla S, Srisim K, Arrayawichanon P, Siritaratiwat W. Concurrent validity of the 10-meter walk test as compared with the 6-minute walk test in patients with spinal cord injury at various levels of ability. Spinal Cord. 2014 Apr;52(4):333-6. doi: 10.1038/sc.2013.171. Epub 2014 Jan 21. PMID 24445972
- [Background] Amatachaya S, Wannapakhe J, Arrayawichanon P, Siritarathiwat W, Wattanapun P. Functional abilities, incidences of complications and falls of patients with spinal cord injury 6 months after discharge. Spinal Cord. 2011 Apr;49(4):520-4. doi: 10.1038/sc.2010.163. Epub 2010 Dec 14. PMID 21151192
- [Background] Baer G, Smith M. The recovery of walking ability and subclassification of stroke. Physiother Res Int. 2001;6(3):135-44. doi: 10.1002/pri.222. PMID 11725595
- [Background] Balasubramanian CK, Bowden MG, Neptune RR, Kautz SA. Relationship between step length asymmetry and walking performance in subjects with chronic hemiparesis. Arch Phys Med Rehabil. 2007 Jan;88(1):43-9. doi: 10.1016/j.apmr.2006.10.004. PMID 17207674
- [Background] Behrman AL, Bowden MG, Nair PM. Neuroplasticity after spinal cord injury and training: an emerging paradigm shift in rehabilitation and walking recovery. Phys Ther. 2006 Oct;86(10):1406-25. doi: 10.2522/ptj.20050212. PMID 17012645
- [Background] Behrman AL, Harkema SJ. Locomotor training after human spinal cord injury: a series of case studies. Phys Ther. 2000 Jul;80(7):688-700. PMID 10869131
- [Background] Bohannon RW. Manual muscle testing: does it meet the standards of an adequate screening test? Clin Rehabil. 2005 Sep;19(6):662-7. doi: 10.1191/0269215505cr873oa. PMID 16180603
- [Background] Bohannon RW, Smith J, Hull D, Palmeri D, Barnhard R. Deficits in lower extremity muscle and gait performance among renal transplant candidates. Arch Phys Med Rehabil. 1995 Jun;76(6):547-51. doi: 10.1016/s0003-9993(95)80509-5. PMID 7763154
- [Background] Brotherton SS, Krause JS, Nietert PJ. A pilot study of factors associated with falls in individuals with incomplete spinal cord injury. J Spinal Cord Med. 2007;30(3):243-50. doi: 10.1080/10790268.2007.11753932. PMID 17684890
- [Background] Brotherton SS, Krause JS, Nietert PJ. Falls in individuals with incomplete spinal cord injury. Spinal Cord. 2007 Jan;45(1):37-40. doi: 10.1038/sj.sc.3101909. Epub 2006 Feb 21. PMID 16491105
- [Background] Calancie B, Needham-Shropshire B, Jacobs P, Willer K, Zych G, Green BA. Involuntary stepping after chronic spinal cord injury. Evidence for a central rhythm generator for locomotion in man. Brain. 1994 Oct;117 ( Pt 5):1143-59. doi: 10.1093/brain/117.5.1143. PMID 7953595
- [Background] Capato TT, Tornai J, Avila P, Barbosa ER, Piemonte ME. Randomized controlled trial protocol: balance training with rhythmical cues to improve and maintain balance control in Parkinson's disease. BMC Neurol. 2015 Sep 7;15:162. doi: 10.1186/s12883-015-0418-x. PMID 26347052
- [Background] Crozier KS, Cheng LL, Graziani V, Zorn G, Herbison G, Ditunno JF Jr. Spinal cord injury: prognosis for ambulation based on quadriceps recovery. Paraplegia. 1992 Nov;30(11):762-7. doi: 10.1038/sc.1992.147. PMID 1484726
- [Background] Dobkin BH. Neuroplasticity. Key to recovery after central nervous system injury. West J Med. 1993 Jul;159(1):56-60. PMID 8351906
- [Background] Graham JE, Ostir GV, Fisher SR, Ottenbacher KJ. Assessing walking speed in clinical research: a systematic review. J Eval Clin Pract. 2008 Aug;14(4):552-62. doi: 10.1111/j.1365-2753.2007.00917.x. Epub 2008 May 2. PMID 18462283
- [Background] Jackson AB, Carnel CT, Ditunno JF, Read MS, Boninger ML, Schmeler MR, Williams SR, Donovan WH; Gait and Ambulation Subcommittee. Outcome measures for gait and ambulation in the spinal cord injury population. J Spinal Cord Med. 2008;31(5):487-99. doi: 10.1080/10790268.2008.11753644. PMID 19086706
- [Background] Lapointe R, Lajoie Y, Serresse O, Barbeau H. Functional community ambulation requirements in incomplete spinal cord injured subjects. Spinal Cord. 2001 Jun;39(6):327-35. doi: 10.1038/sj.sc.3101167. PMID 11438855
- [Background] Lord SR, Murray SM, Chapman K, Munro B, Tiedemann A. Sit-to-stand performance depends on sensation, speed, balance, and psychological status in addition to strength in older people. J Gerontol A Biol Sci Med Sci. 2002 Aug;57(8):M539-43. doi: 10.1093/gerona/57.8.m539. PMID 12145369
- [Background] Pang MY, Yang JF. The initiation of the swing phase in human infant stepping: importance of hip position and leg loading. J Physiol. 2000 Oct 15;528 Pt 2(Pt 2):389-404. doi: 10.1111/j.1469-7793.2000.00389.x. PMID 11034628
- [Background] Wirz M, van Hedel HJ, Rupp R, Curt A, Dietz V. Muscle force and gait performance: relationships after spinal cord injury. Arch Phys Med Rehabil. 2006 Sep;87(9):1218-22. doi: 10.1016/j.apmr.2006.05.024. PMID 16935058